CLINICAL TRIAL: NCT06476873
Title: Substance Use Disorder in Chemsex Practice: Evaluation of the Prevalence of the Disorder Among Users Via an Online Self-questionnaire
Brief Title: Substance Use Disorder in Chemsex Practice
Acronym: TU CHEMSEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A00737-40
Record Dates: First submitted 2024-06-17; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Addiction Chemical; Use, Substance
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Online self-questionnaire. — Descriptive, cross-sectional study This study is aimed at adult chemsex users over the last 12 months (having experimented with chemsex at least once over the last 12 months) and with a good understanding of French.
  An online LimeSurvey-type self-questionnaire will be accessible via a URL link to collect and secure the data. A presentation of the study, information on chemsex and help and care services, as well as the information note will be available.
  The questionnaire will be distributed via a QR code, giving direct access to the study's web page, or directly via the web link. Posters and flyers will be used in hospitals and/or private clinics, addictology centers, STI prevention and screening centers and associations, as well as via social networks, dating apps and sites, and the online and print press.

SUMMARY:
The main aim of this descriptive cross-sectional study is to assess the prevalence of chemsex substance use disorder among chemsexers via an online self-questionnaire.

DETAILED DESCRIPTION:
Chemsex appeared in Europe around 2006 and in France in 2010. It involves the use of psychoactive substances in a sexual context to enhance, initiate, facilitate or prolong sexual intercourse through the psychoactive effects of the molecules consumed. These molecules are essentially synthetic cathinones, GHB/GBL, MDMA, methamphetamines, cocaine and ketamine. These products are often used in combination with erectile dysfunction treatments (side effects of the molecules). This practice is thought to affect almost 20% of MSM.

This use has numerous social, somatic, psychiatric and addictive consequences. Studies have mainly focused on infectious risks, psychiatric complications (e.g. anxiety and depression) or the prevalence of this phenomenon. However, no study has assessed the prevalence of chemsex-related substance use disorders among these users.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Proficiency in written French
* Have practised chemsex at least once in the last 12 months.
* Agree to participate in the study.

Exclusion Criteria:

* Have not experimented with chemsex in the last 12 months
* Participation in other ongoing research
* Insufficient written comprehension of French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
DSM-5 diagnosis of substance use disorder for chemsex. | 1 day
  Assessment of the prevalence of chemsex substance use disorder among chemsexers via an online self-questionnaire.

SECONDARY OUTCOMES:
Describing the sociodemographic characteristics of this population | 1 day
  Socio-demographic characteristics
Describing the consumption practices of this population | 1 day
  Consumption practices
Describing the sexual practices of this population | 1 day
  Sexual practices
Explore the existence of chemsex use disorder as a clinical entity in its own right | 1 day
  DSM-5 diagnostic criteria for substance use disorder, adapted to assess chemsex addiction as a single clinical entity

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Charles PERRENS, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diestelmann M, Zangl A, Herrle I, Koch E, Graw M, Paul LD. MDPV in forensic routine cases: Psychotic and aggressive behavior in relation to plasma concentrations. Forensic Sci Int. 2018 Feb;283:72-84. doi: 10.1016/j.forsciint.2017.12.003. Epub 2017 Dec 8. PMID 29275216
- [Background] Blanc JV, Burdairon JD, Malandain L, Ferreri F, Mouchabac S, Adrien V. Attachment and Mental Health of Men Having Sex with Men Engaging in Chemsex: Is Substance Abuse Only the Tip of the Iceberg? J Homosex. 2024 Oct 14;71(12):2875-2894. doi: 10.1080/00918369.2023.2266086. Epub 2023 Oct 10. PMID 37815854
- [Background] Serre A, Vuillot O, Eiden C, Gambier J, Berger A, Mathieu O, Nefau T, Sebbane M, Donnadieu-Rigole H, Peyriere H. Acute Psychiatric Disorders Related to Fake Cathinone: Ephylone. J Anal Toxicol. 2019 Aug 23;43(7):e1-e2. doi: 10.1093/jat/bkz020. No abstract available. PMID 31095710
- [Background] Evers YJ, Van Liere GAFS, Hoebe CJPA, Dukers-Muijrers NHTM. Chemsex among men who have sex with men living outside major cities and associations with sexually transmitted infections: A cross-sectional study in the Netherlands. PLoS One. 2019 May 14;14(5):e0216732. doi: 10.1371/journal.pone.0216732. eCollection 2019. PMID 31086390
- [Background] Gilbart VL, Simms I, Gobin M, Oliver I, Hughes G. High-risk drug practices in men who have sex with men. Lancet. 2013 Apr 20;381(9875):1358-1359. doi: 10.1016/S0140-6736(13)60882-X. No abstract available. PMID 23601946